CLINICAL TRIAL: NCT07230145
Title: A Double-Blind, Randomized, Dose-Escalating Phase I Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single-Dose SHR-4658 in Healthy Volunteers or Volunteers With Elevated Blood Pressure
Brief Title: A Trial of SHR-4658 in Healthy Volunteers or Volunteers With Elevated Blood Pressure
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Suncadia Pharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-4658-101
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-4658 Group (Experimental)
  Interventions: Drug: SHR-4658 Injection.
- SHR-4658 Placebo Group (Placebo Comparator)
  Interventions: Drug: SHR-4658 Placebo Injection

INTERVENTIONS:
Drug: SHR-4658 Injection. — SHR-4658 injection.
  Arms: SHR-4658 Group
Drug: SHR-4658 Placebo Injection — SHR-4658 placebo injection.
  Arms: SHR-4658 Placebo Group

SUMMARY:
This is a clinical study to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamic and immunogenicity of single subcutaneous injection of SHR-4658 in healthy volunteers and volunteers with elevated blood pressure.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent.
2. Blood pressure as defined in the protocol.
3. Male or female，aged 18 to 55 years (inclusive).
4. Meet the weight standard.

Exclusion Criteria:

1. Known history or current clinically significant disease.
2. Protocol-defined risk factors for disease.
3. Participated in clinical trials of other drugs or medical devices.
4. Pregnant or nursing women.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs) | Approximately 16 weeks.

SECONDARY OUTCOMES:
Area under the concentration-time curve from time 0 to the last time point (AUC0-last) | Approximately 16 weeks.
Area under the concentration-time curve from time 0 to infinity (AUC0-inf) | Approximately 16 weeks.
Maximum observed concentration (Cmax) | Approximately 16 weeks.
Time to maximum observed concentration (Tmax) | Approximately 16 weeks.
Apparent clearance (CL/F) | Approximately 16 weeks.
Apparent volume of distribution (Vd/F) | Approximately 16 weeks.
Terminal elimination half-life (t1/2) | Approximately 16 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided